CLINICAL TRIAL: NCT07138352
Title: An Open-label, Single-center, Randomized, Two-treatment, Two-period, Two-sequence, Single Dose, Crossover Study to Evaluate the Oral Comparative Bioavailability of XS003 (Nilotinib) Capsules 192 mg Under Fasted and Fed Conditions in Healthy, Adult Subjects.
Brief Title: Bioavailability Study of XS003 (Nilotinib)
Acronym: XS003-14
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xspray Pharma AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: XS003-14
Record Dates: First submitted 2025-07-29; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a single-dose, open-label, randomized, crossover study to evaluate the comparative oral bioavailability of XS003 (nilotinib) Capsules 192 mg (4X 48 mg) of Xspray Pharma AB, Sweden under fasted conditions comparing with XS003 (nilotinib) Capsules 192 mg (4X 48 mg) of Xspray Pharma AB, Sweden in healthy, adult, human subjects under fed conditions.
Masking Description: N/A as it is an open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- XS003 fasted condition (Experimental): XS003 (nilotinib) Capsules 192 mg (4X 48 mg) under fasted conditions.
  Interventions: Drug: XS003 under fed and fasted condition
- XS003 fed condition (Experimental): XS003 (nilotinib) Capsules 192 mg (4X 48 mg) under fed conditions
  Interventions: Drug: XS003 under fed and fasted condition

INTERVENTIONS:
Drug: XS003 under fed and fasted condition — XS003 under fed and fasted condition

SUMMARY:
An open label, single-center, randomized, two-treatment, two-period, two-sequence, single dose, crossover, study under fasted and fed conditions.

DETAILED DESCRIPTION:
This is a single-dose, open-label, randomized, crossover study to evaluate the comparative oral bioavailability of XS003 (nilotinib) Capsules 192 mg (4X 48 mg) of Xspray Pharma AB, Sweden under fasted conditions comparing with XS003 (nilotinib) Capsules 192 mg (4X 48 mg) of Xspray Pharma AB, Sweden in healthy, adult, human subjects under fed conditions.

This will enroll up to 48 healthy, adult, human subjects. Each sequence will enroll 24 healthy, adult, human subjects. There will be at least 10 days between each drug administration.

Adverse events will be recorded from the signing of ICF throughout the study. In each period, the subjects will be housed for approximately 14 hours before and at least 24 hours after the drug administration. Subjects will return to clinical facility for ambulatory samples at 48.00, 72.00, 96.00 and 120.00 hours post dose.

ELIGIBILITY:
Inclusion Criteria:

* A willing study participant to become eligible for the study must fulfil all of the below inclusion criteria.
* Healthy, human beings 18 and 55 years of age inclusive at the time of screening.
* Subjects, having a body mass index between ≥18.0 kg/m2 and <32.0 kg/m2.
* Subjects must be able to provide written informed consent.
* Acceptable medical history, physical examination, ECG, laboratory investigations per the Investigator.
* Female subjects must meet at least one of the following requirements:

  * Agree to abstain from sexual intercourse from screening, throughout the duration of the study and for at least 90 days after the last study drug administration.
  * Have used and agree to continue to use a reliable method of contraception (e.g., hormonal contraceptives, condom with spermicide, IUD) for at least 30 days before initial dosing, throughout the duration of the study and for at least 90 days after the last study drug administration.
  * Surgically sterile (bilateral oophorectomy or hysterectomy, bilateral tubal ligation at least 3 months before initial dosing or Essure® device placement).
  * At least 1 year postmenopausal and have a documented FSH level ≥ 40 mIU/mL at screening.
* Male subjects who are not surgically sterile must agree to abstain from sexual intercourse (complete abstinence) or use appropriate contraceptive measures and agree to not impregnate a female partner(s) and not to donate sperm throughout the entire study, including the washout periods, and for at least 90 days after the last study drug administration. Examples of acceptable methods of contraception include a double-barrier method of contraception (e.g., condom with spermicide). Other forms of contraception may be acceptable, at the discretion of the Investigator.
* Clinical laboratory values should be within the laboratory's stated normal range. If not within this range, they must be without clinical significance, as determined by the Investigator (with the exception of those labs specifically listed in Section 9.2.).
* The subject is able to communicate meaningfully with study personnel and is anticipated to be able to comply fully with study procedures and must be willing and able to communicate and participate in the whole study.
* Male subjects should not donate sperm during the study and for 90 days after the last administration of IMP.

Exclusion Criteria:

* A willing study participant will be excluded from the study, if any of the below criteria is met.
* Systolic blood pressure is less than 100 mm of Hg or more than 140 mm of Hg.
* Diastolic blood pressure is less than 60 mm of Hg or more than 90 mm of Hg.
* Note: If vital signs are out-of-range, the investigator may obtain one additional reading so that up to 2 consecutive assessments are made within 1.00 hour with the subject seated quietly during the 5 minutes preceding the assessment.
* Body temperature less than 95.0 °F (35.0 °C) or more than 98.6°F (37.0°C).
* Heart rate less than 60/min or more than 100/min.
* History of hypersensitivity or idiosyncratic reaction to investigational drug product or any other related drugs.
* History of malignancy, cardiovascular, pulmonary, hepatic, renal, gastrointestinal, endocrine, immunological, dermatological, neurological, or psychiatric disease or disorder considered clinically significant in the opinion of the Investigator.
* Taken drugs that are substrates or inhibitors of P-glycoproteins in last 30 days prior to the check-in.
* History of hematological, malignant, and bleeding disorders.
* On anticoagulant therapy, within 4 weeks prior to the check-in.
* History of hypokalemia, hypomagnesemia, or a history of cardiac disease.
* History of cholecystectomy or gall stones.
* History of any drug or alcohol abuse in the past 2 years.
* History of intake of strong CYP3A4 inhibitors (see Table 5) or inducers within 4 weeks prior to the check-in.
* History of intake of drugs known to prolong the QTc interval within 4 weeks prior to the check-in
* History of rare hereditary problems of galactose intolerance, severe lactase deficiency with a severe degree of intolerance to lactose-containing products, or of glucose- galactose malabsorption.
* A prolonged QTc interval (QTcF greater than 450 msec demonstrated on ECG at Screening.)
* Any clinically significant ECG abnormalities that, in the Investigator's opinion, would compromise the subject's safety.
* History or family history of long QT syndrome.
* Significant history or current evidence of risk factors for Torsade de Pointes (TdP).
* History of Gilbert syndrome.
* Having poor vein access.
* Male subjects with pregnant or breastfeeding partners.
* Taking, or have taken, any prescribed or over-the-counter drug or herbal remedies, vitamins, or minerals and intake of any medication except caffeine, ranitidine, paracetamol, diclofenac sodium and ondansetron within 14 days before check-in (other than up to 4 g of paracetamol/acetaminophen per day).
* Consumption of xanthine containing food or beverages (like tea, coffee, chocolates, and flavored drinks) within 48 hours before check-in of each period.
* Consumption of grapefruit or grapefruit juice, pomegranate, or pomegranate juice, pomelo, starfruit, Seville oranges and St. John's Wort within 14 days before check-in.
* Consumption of tobacco containing products (including smoking cigarettes or chewing tobacco products), e-cigarettes and/or nicotine replacement products within 3 months before check-in.
* Consumption of alcoholic beverages within 48 hours before check-in.
* Positive drugs of abuse screen at Screening or upon check-in of any period. Based on local regulations, if positive for tetrahydrocannabinol, evaluation will be performed by the PI based on last usage date (must be at least 14 days prior to the initial dosing and throughout the duration of the entire study period).
* Positive alcohol (breath or urine) test screen at screening or upon check-in of any period.
* Positive urine cotinine test screen at screening or upon check-in of any period.
* Participated in any other clinical study or donated blood within 30 days before check-in.
* Positive screens for serum Hepatitis B virus surface antigen (HBsAg), Hepatitis C virus antibody ( HCV Ab) or Human Immunodeficiency Virus (HIV-1 & 2).
* Participated in contact sports or unaccustomed strenuous exercise within 72 hours before check-in of any period.
* History of clinically significant allergy or any allergy or sensitivity to nilotinib, or history of any food or drug hypersensitivity or intolerance which, in the opinion of the Investigator, would compromise the safety of the subject or the study.
* Significant history or current evidence of chronic infectious disease, system disorders, organ dysfunction especially cardiovascular disorders (e.g., arterial vascular occlusive events), respiratory disorders, renal or hepatic disorders, diabetes, or obesity.
* Subjects with greater than the safety laboratory upper limit of normal values of ALP, ALT, AST and total bilirubin.
* Estimated glomerular filtration rate (eGFR) < 90 mL/min at screening
* Subjects with less than the safety laboratory lower limit of normal values for potassium or magnesium.
* Clinically significant history or presence of gastrointestinal disease or history of malabsorption within the last year, as determined by the Investigator.
* Positive pregnancy test (for females) at screening or upon check-in of any period.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2024-10-03 (Actual); Primary Completion 2025-01-08 (Actual); Study Completion 2025-01-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the comparative bioavailability Cmax of XS003 (nilotinib) Capsules 192 mg (4X 48 mg) under fasted and fed conditions in healthy, adult, human subjects. | PK samples will be collected at pre-dose (0.00) and between 0.50 and 120.00 hours post dose
  Primary PK endpoints: Cmax: Maximum measured analyte concentration in the biological fluid.
To evaluate the comparative bioavailability AUC of XS003 (nilotinib) Capsules 192 mg (4X 48 mg) under fasted and fed conditions in healthy, adult, human subjects. | PK samples will be collected at pre-dose (0.00) and between 0.50 and 120.00 hours post dose
  Primary PK endpoints: AUC0-t: Time of the maximum observed drug concentration.

SECONDARY OUTCOMES:
To evaluate the safety (adverse events (AE)) of XS003 (nilotinib) Capsules 192 mg (4X 48 mg) under fasted and fed conditions in healthy, adult, human subjects. | From Screening until end of study, i.e. up to 56days
  To collect data on treatment related and non treatment related adverse events as assessed by CTCAE v4.0"
To evaluate the safety and tolerability (ECG, elektrocardiogram) of XS003 (nilotinib) Capsules 192 mg (4X 48 mg) under fasted and fed conditions in healthy, adult, human subjects. | From Screening until end of study, i.e. up to 56days
  Safety variables collection will include ECG, elektrocardiogram QT Interval

CONTACTS AND LOCATIONS:
Overall Officials: Maria Klockare, Study Director — Xspray Pharma
Locations (1):
- QPS Missouri, Springfield, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
This is an Bioavailibility study so IPD is N/A